CLINICAL TRIAL: NCT06176248
Title: Evaluation of the Efficacy of Suprascapular Nerve Block in Adhesive Capsulitis: a Randomized Controlled Superiority Trial
Brief Title: Evaluation of the Efficacy of Suprascapular Nerve Block in Adhesive Capsulitis
Acronym: BAC-Reims
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PA23085*
Record Dates: First submitted 2023-07-24; First posted 2023-12-19 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Adhesive Capsulitis
MeSH Terms: conditions — Bursitis | interventions — Triamcinolone Acetonide; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Block and arthrodistension (Active Comparator)
  Interventions: Drug: Triamcinolone Acetonide
- Placebo and arthrodistension (Placebo Comparator)
  Interventions: Drug: saline solution

INTERVENTIONS:
Drug: Triamcinolone Acetonide — 1 injection of local anaesthetic (5 ml levobupivacaine 2.5 mg/mL) opposite the subscapular nerve, under ultrasound control, in a lateral decubitus or sitting position. Subsequently, they underwent Xray-controlled arthrodistension by injection of 1 ml of Triamcinolone Acetonide, combined with 10 ml of visipaque 270 contrast medium and 5 ml of Xylocaine.
  Arms: Block and arthrodistension
Drug: saline solution — intramuscular injection of 1 ml saline under ultrasound control under the same conditions as the experimental group. Subsequently, they will undergo Xray-controlled arthrodistension under the same conditions as the experimental group
  Arms: Placebo and arthrodistension

SUMMARY:
This is a double-blind interventional superiority study evaluating the efficacy of suprascapular nerve block in addition to conventional therapies for adhesive capsulitis.

Adhesive capsulitis is a pathology that results in reduced shoulder mobility due to retraction of the periarticular capsule. It may be primary or secondary to traumatic or neurological events, or associated with diabetes in particular.

The usual treatment includes re-education sessions to improve joint amplitude and restore shoulder mobility. In persistent forms, intra-articular injection of cortisone is combined with distension of the capsule with a local anaesthetic under radiographic control.

In some countries, subscapular nerve block (reversible anaesthesia) is used to improve pain. The combination of arthrodistension and subscapular nerve block has never been performed to accelerate the healing process.

The aim of this study is to compare the performance of these two procedures together against the reference technique alone on time to improvement with the number of patients improved at one month according to the Constant score.

This score is used to assess shoulder pain and function, with a significant improvement above eight points.

DETAILED DESCRIPTION:
The glenohumeral joint is a highly mobile joint involving abduction, anterior elevation, external rotation and internal rotation. It is composed of a capsule innervated by the suprascapular nerve. Retractile capsulitis is a frequent pathology, affecting 2 to 5% of the general population, and associating both pain and stiffening of the joint, leading to functional discomfort, particularly in abduction and external rotation movements. It is due to capsular retraction of the shoulder joint, which may be idiopathic or secondary to traumatic or neurological etiology, or associated with diabetes. In the majority of cases, this pathology leads to recovery, but the time to total recovery is variable, ranging from six months to one year. Some studies have even shown the persistence of symptoms, with an average follow-up time of four years in some patients. The majority of patients are off work due to the functional discomfort associated with shoulder stiffness.

Therapeutic management is currently poorly codified. Physiotherapy using active mobilization maneuvers has been shown to improve joint amplitudes, and is used as a first-line treatment. In the event of persistent symptoms, cortisone infiltration has been evaluated using a variety of protocols, including sub-acromial and intra-articular infiltration, as well as arthro-distension, which consists of dilating the capsule under radiological control using 1 intra-articular injection of xylocaine, corticoids and contrast medium. In France, arthrodistension has become the reference technique, as it is more effective than intra-articular infiltration of cortisone derivatives. In fact, several trials and meta-analyses have demonstrated short-term superiority in improving the pain associated with capsulitis and, above all, better progress in terms of joint amplitude, as assessed in particular by Constant's algo-functional scores.

If adhesive capsulitis persists despite these therapies, arthroscopic surgery is sometimes performed.

The suprascapular nerve is a mixed nerve whose sensitive component is the main sensitive branch innervating the shoulder. An anaesthetic block of this nerve provides a punctual reduction in painful sensations in the shoulder, enabling less painful arthrodistension and pain-free physiotherapy sessions for faster joint amplitude work. Several studies have compared suprascapular nerve block versus intra-articular infiltration in this condition, with conflicting results which nevertheless show a trend towards improved joint amplitudes and earlier onset of pain in the anesthetic block group. However, no study has compared suprascapular nerve block with arthrodistension, which remains the standard treatment in Europe. Moreover, no study has investigated the superiority of adding this therapy to arthrodistension. Our hypothesis is that suprascapular nerve block combined with arthrodistension may accelerate healing.

The main benefit expected for the patient is the shortening of the time to improvement (recovery of joint amplitudes, functional improvement and improvement in quality of life).

The expected benefits for society would be to improve therapeutic management and reduce healthcare consumption and indirect costs (time off work).

The foreseeable risks are low, with a risk of allergy to the anesthetic and a transient motor deficit (4h) in the supra-scapular nerve territory.

ELIGIBILITY:
Inclusion Criteria:

* Patient treated for adhesive capsulitis corresponding to a loss of passive amplitude of more than 20° in external rotation elbow to body and/or abduction in relation to the contralateral shoulder.
* Patient over 18 years of age
* Patient covered by a social security scheme
* Presence of an accompanying person on the day of the procedure for the return trip
* Patient having signed the consent form to participate in the study

Exclusion Criteria:

* Patient protected by law
* Pregnant women
* Patient who has had shoulder surgery less than six months old
* Patient unable to undergo rehabilitation within one month of surgery
* Allergy to one of the products used (anesthetic, iodinated contrast medium)
* Neuro-orthopedic disorder hampering clinical recovery
* Hemostasis disorder contraindicating block (no discontinuation of anticoagulants according to SFAR recommendations, congenital hemostasis disorder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2027-01-11 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Constant score | 1 month
  The Constant score measured at inclusion and at 1 month in both groups. Calculation of the difference in score between the two times (minimum 0 - maxumum 100)

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: No